CLINICAL TRIAL: NCT06074133
Title: A Combined Biomarker Model for Risk Stratification of Indeterminate Pulmonary Nodules A Multicenter Prospective Observational Pilot Study
Brief Title: A Combined Biomarker Model for Risk Stratification of Indeterminate Pulmonary Nodules
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric Grogan, Professor of Thoracic Surgery & Medicine, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC-EDTHO23230; NCI-2023-05725 (Registry Identifier: NCI, Clinical Trials Reporting Program); 5R01CA252964-02 (NIH)
Record Dates: First submitted 2023-09-19; First posted 2023-10-10 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Nodule
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indeterminate Pulmonary Nodules: A combined biomarker model (hs-CYFRA 21-1, radiomics, Mayo) score will be obtained to estimate potential clinical utility compared to the Mayo Model.
  Interventions: Procedure: Blood collection; Procedure: Chest Computed Tomography

INTERVENTIONS:
Procedure: Blood collection — Undergo blood draw
Procedure: Chest Computed Tomography — Undergo standard of care chest Computed Tomography

SUMMARY:
This is a prospective, multicenter observational study aim at estimating the potential clinical utility of the CBM and at establishing the SOPs and protocols for a future randomized control trial.

DETAILED DESCRIPTION:
Objectives:

* To obtain the combined biomarker model (hs-CYFRA 21-1, radiomics, Mayo) score in a prospective observational trial and estimate potential clinical utility compared to the Mayo Model.
* To establish standard operating procedures (SOPs) and protocols in a prospective observational trial in anticipation of a future randomized control trial. These include the REDCAP data input protocols, the radiomic protocols, blood draws in the CLIA environment, and estimating the CBM score in a time reasonable for clinical practice (< 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Adults > 21 y/o
* IPNs 8-30mm referred for evaluation Figure 4. AUC and reclassification of Combined Biomarker Model
* Intermediate risk IPN defined as 10-70% risk after applying Mayo risk predictor model
* Solid nodules or part-solid nodules with solid component >=8mm
* CT scan with nodule of concern performed within 60 days of enrollment

Exclusion Criteria:

Pure ground glass nodule or subsolid nodule with solid component <8mm

* Currently on therapy for any cancer
* History of primary lung cancer within the last 5 years
* Multiple nodules highly suspicious for metastatic disease
* Other malignancy within the last 2 year - Excluding skin cancer other than melanoma
* Pregnant women
* Prisoners
* Inability to provide informed consent
* Serologic evidence of active fungal infection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from pulmonary or thoracic clinics that have indeterminate pulmonary nodules
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with benign disease who underwent invasive diagnostic procedures. | Up to approximately 2 years
The time to diagnosis (in days) for patients with cancer. | Up to approximately 2 years
Measure time needed to provide the CBM Value to clinician | Up to approximately 2 years
  Number of days
Measure time needed to obtain hs CYFRA 21-1 values | Up to approximately 2 years
  Number of hours (days)
Measure time needed to perform radiomics | Up to approximately 2 years
  Number of hours (days)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Grogan, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (4):
- United States (4):
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - VA Tennessee Valley Healthcare Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT06074133/ICF_000.pdf